CLINICAL TRIAL: NCT07236320
Title: Neoadjuvant Immunochemotherapy Versus Chemoradiotherapy in Locally Advanced Esophageal Cancer: A Real-World Study
Brief Title: Neoadjuvant Immunochemotherapy vs Chemoradiotherapy in ESCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Chief Surgeon / Professor, Department of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCH-TS2503
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICT group (Experimental)
  Interventions: Drug: Neoadjuvant immunochemotherapy
- NCRT group (Active Comparator)
  Interventions: Drug: Neoadjuvant Chemoradiotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — NACI group patients received treatment of minimally 2 cycles of ICIs agent (mainly camrelizumab or toripalimab, 200 mg every 3 weeks (200 mg every 3 weeks)) combined with concurrent chemotherapy.
  Arms: NICT group
Drug: Neoadjuvant Chemoradiotherapy — NCRT group patients followed the concurrent NCRT treatment, and the total neoadjuvant radiotherapy dose was 40.0-50.4Gy with 1.8-2.14 Gy fractions and 5 fractions/week.
  Arms: NCRT group

SUMMARY:
This retrospective real-world study aimed to compare neoadjuvant immunochemotherapy (NICT) and neoadjuvant chemoradiotherapy (NCRT) followed by esophagectomy in patients with locally advanced esophageal squamous cell carcinoma (ESCC). A total of 203 consecutive patients treated at Sichuan Cancer Hospital between March 2018 and March 2022 were analyzed (NICT: 59; NCRT: 144). The primary endpoints were overall survival (OS) and disease-free survival (DFS); secondary endpoints included pathological complete response (pCR), tumor regression grade (TRG), and R0 resection rate. After inverse probability of treatment weighting adjustment, baseline characteristics were balanced between groups. Both groups achieved comparable long-term OS and DFS, while NCRT showed higher rates of local pathological response. Exploratory subgroup analysis suggested that patients achieving pCR after NICT might have superior survival outcomes. The study indicates that NICT provides similar long-term survival compared to NCRT and may offer immunologic advantages for selected responders, warranting further validation in prospective multicenter trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Histologically confirmed thoracic ESCC
* Clinical stage cT1N+M0 or cT2-4aN0-3M0
* Received neoadjuvant therapy (immunochemotherapy or chemoradiotherapy) followed by esophagectomy

Exclusion Criteria:

* History of other malignancies
* Did not complete neoadjuvant therapy or required salvage surgery
* Incomplete baseline or follow-up data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Time from first treatment to death from any cause or last follow-up.
Disease-Free Survival (DFS) | 5 years
  Time from surgery to recurrence, death, or last follow-up.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) rate | 3 months
Tumor Regression Grade (TRG) | 3 months
R0 resection rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared because this is a retrospective study based on patient medical records, and the data contain potentially identifiable clinical information. Ethical approval for this study was granted under the condition that data would be used only for internal analysis at Sichuan Cancer Hospital & Institute. De-identified summary-level results are provided within the publication.